CLINICAL TRIAL: NCT04716426
Title: Use of APT™ T3X to Decrease the COVID-19 Contamination Rate in Humans
Brief Title: APT™ T3X on the COVID-19 Contamination Rate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Collaborators: Santa Casa de Porto Alegre (Other)
Responsible Party: Principal Investigator, Ernesto Cesar Pinto Leal Junior, Full professor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 4.485.847
Record Dates: First submitted 2021-01-18; First posted 2021-01-20 (Actual); Results first posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: COVID-19
Keywords: Prevention; Tetracycline hydrochloride; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A participating researcher not involved in the recruitment and evaluation of the volunteers will carry out the randomization process. This researcher will be instructed not to disclose the randomization codes in the intervention groups to any of the volunteers and to the other researchers involved in the study, until its completion. The intervention bottles will be exactly the same regardless of whether it is APT™ T3X or placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tetracycline hydrochloride 3% (Experimental): 4 drops of tetracycline hydrochloride 3% (APT™ T3X) applied inside of the nasal channels and inside of nostrils, once a day, every day for 21 days (except health professionals that will be instructed to use 4 drops of APT™ T3X twice a day, every day for 21 days.
  Interventions: Drug: Tetracycline hydrochloride 3%
- Placebo (Placebo Comparator): 4 drops of placebo applied inside of the nasal channels and inside of nostrils, once a day, every day for 21 days (except health professionals that will be instructed to use 4 drops of APT™ T3X twice a day, every day for 21 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tetracycline hydrochloride 3% — Proprietary formulation composed of FDA approved inactive ingredients and the active pharmaceutical ingredient tetracycline hydrochloride.
  Other Names: APT™T3X
  Arms: Tetracycline hydrochloride 3%
Drug: Placebo — Formulation composed of FDA approved inactive ingredients.
  Arms: Placebo

SUMMARY:
The new coronavirus 2019 (COVID-19) was declared a pandemic by the World Health Organization (WHO), due to the alarming levels of spread, severity and inaction. Dealing with COVID-19 must be done on different fronts, such as mitigation, treatment and prevention. Therefore, strategies and therapies that can help reduce the COVID-19 rate of contamination are still important alternatives at this time of the pandemic.

The Advanced Penetration Technology™ (APT™) is intellectual property owned by Patient Focused Tele-Health, LLC, a Rockwall, Texas based company. The company's focus is improving over-the-counter (OTC) topical formulations, allowing consumers better therapeutic outcomes with non-prescription medications.

The Advanced Penetration Technology™ (APT™) is a patent-pending, proprietary transdermal dual carrier formulation. This formulation provides improved dermal penetration and efficacy of topical API's. Additionally, the APT™ imparts both a mechanical and biochemical effect on the microbe/fungal cell walls providing a highly effective method of destruction of microbes. These unique properties impart the broad spectrum anti-viral capability to the APT™ Tetracycline 3% formulation, breaking barriers in pharmacology and virology.

The topical formulation APT™ Tetracycline 3% formulation (APT ™ T3X), is a FDA registered, Non-Prescription product. This formulation is used in an off label manner as an intranasal application for prevention of COVID-19 and other viruses. The APT™ T3X as a topical application will penetrate through and into the mucus layer and deeper. This barrier of coverage will provide a mitigation effect to decrease the viral load of exposure and infection. The efficacy of APT™ T3X is due to disrupting the lipid envelope in seconds, hence neutralizing the virus.

Previous tests were performed with APT™ T3X and the results found were promising. However, these tests were performed only in vitro and clinical studies demonstrating the ability of the APT™ T3X to decrease viral exposure and contamination by COVID-19 are necessary to confirm the possible prophylactic effect, allowing the formulation to be widely distributed to the general population.

Therefore, the aim of this project is to evaluate the efficacy of the APT™ T3X compared to placebo to decrease COVID-19 contamination rate in humans.

DETAILED DESCRIPTION:
To achieve the proposed objective it will be performed a randomized, triple blind, placebo-controlled trial. The volunteers will be randomly allocated to two intervention groups: APT™ T3X or placebo. The volunteers will be blinded to the treatment received.

One hundred volunteers will be recruited for the study (50 volunteers per group). As this is a preliminary study, the number of volunteers was determined by a convenience sample.

The volunteers randomly allocated to the two groups will be instructed to use the APT™ T3X or placebo, once a day, every day for 21 days (except health professionals that will be instructed to use APT™ T3X or placebo twice a day, every day for 21 days).

All data will be collected by a blinded assessor. The investigators will analyze:

1. COVID-19 contamination rate.
2. Presence of adverse events.
3. Number of adverse events.
4. Frequency of adverse events.
5. Other virus or bacteria contamination rate.

Statistical analysis: The results obtained will first be tested for normality using the Kolmogorov-Smirnov test. The chi-square test or Fisher's exact test for two independent proportions will be used in the statistical analysis of the primary outcome of this study, the COVID-19 contamination rate and for the secondary outcomes: presence of adverse events and other virus or bacteria contamination rate. For the other secondary outcomes, the number of adverse events and frequency of adverse events, the Wilcoxon test will be used if this outcome does not present a normal distribution. If this outcome presents a normal distribution, the two-tailed, unpaired t test will be used. The level of significance used will be 5% (p <0.05).

ELIGIBILITY:
Inclusion Criteria:

* good general health (without serious health problems);
* tested negative, by means of immunoglobulin (Ig) G and IgM serology tests and chain real-time polymerase chain reaction (RT-PCR), for COVID-19.

Exclusion Criteria:

* previous immunization against COVID-19;
* allergy to tetracycline hydrochloride;
* diagnosis of Lyme disease;
* immunocompromised;
* share housing with someone diagnosed with COVID-19 at the time of the baseline evaluation;
* serious illnesses, such as cancer, kidney failure, decompensated cardiorespiratory and metabolic diseases, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-01-28 (Actual); Primary Completion 2021-03-25 (Actual); Study Completion 2021-03-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Santa Casa de Misericórdia de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was performed between January 28, 2021 and March 25, 2021. The volunteers were recruited at Santa Casa de Misericórdia de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil.
Period: Overall Study
Arm/Group | Tetracycline Hydrochloride 3% | Placebo
Started | 50 | 50
Completed | 48 | 49
Not Completed | 2 | 1
Not completed — Vaccination | 1 | 1
Not completed — Contamination | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tetracycline Hydrochloride 3% | Placebo | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.96 (13.66) | 43.10 (13.49) | 41.03 (13.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 23 | 50
  Male | 23 | 27 | 50
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Brazil | 50 | 50 | 100
Height [Mean (Standard Deviation); unit: cm] | 169 (8) | 169 (10) | 169 (9.30)
Weight [Mean (Standard Deviation); unit: Kg] | 78.55 (14.81) | 78.68 (15.69) | 78.62 (15.19)
Comorbidities [Number; unit: participants] | 14 | 13 | 27

OUTCOME MEASURES:

1. Primary Outcome: COVID-19 Contamination Rate.
Description: Rate of how many people were infected with COVID-19 over the course of the study in each group.
Time Frame: 22 days after randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Tetracycline Hydrochloride 3% | Placebo
Number analyzed (Participants) | 50 | 50
Participants | 2 | 5

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Number of participants who presented adverse events.
Time Frame: 22 days after randomization.
Measure: Number; unit: participants
Arm/Group | Tetracycline Hydrochloride 3% | Placebo
Number analyzed (Participants) | 50 | 50
participants | 17 | 23

3. Secondary Outcome: Average Number of Adverse Events
Description: Average number of adverse events over the course of the study.
Time Frame: 22 days after randomization.
Measure: Mean (Standard Deviation); unit: adverse events
Arm/Group | Tetracycline Hydrochloride 3% | Placebo
Number analyzed (Participants) | 50 | 50
adverse events | 0.65 (1.11) | 0.94 (1.25)

4. Secondary Outcome: Days Over Which an Adverse Event Was Reported
Description: Average days over which an adverse event was reported.
Time Frame: 22 days after randomization.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Tetracycline Hydrochloride 3% | Placebo
Number analyzed (Participants) | 50 | 50
Days | 0.36 (2.2) | 0.28 (1.67)

5. Secondary Outcome: Other Virus or Bacteria Contamination Rate.
Description: Rate of how many people were infected with influenza or pneumonia over the course of the study in each group.
Time Frame: 22 days after randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Tetracycline Hydrochloride 3% | Placebo
Number analyzed (Participants) | 50 | 50
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 22 days
Description: The adverse events were collected through a diary filled by the volunteers during the trial.
Arm/Group | Tetracycline Hydrochloride 3% | Placebo
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 17/50 | 23/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tetracycline Hydrochloride 3% (N=50) | Placebo (N=50)
Itch (Respiratory, thoracic and mediastinal disorders) | 5 (46) | 4 (17)
Coryza (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 4 (25)
Sneeze (Respiratory, thoracic and mediastinal disorders) | 11 (84) | 12 (35)
Nasal irritation (Respiratory, thoracic and mediastinal disorders) | 2 (26) | 4 (25)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (15)
Shed tears (Eye disorders) | 5 (60) | 4 (31)
Nasal burning (Respiratory, thoracic and mediastinal disorders) | 4 (24) | 7 (32)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (8)
Earache (Ear and labyrinth disorders) | 1 (2) | 0 (0)
Nosebleed (Injury, poisoning and procedural complications) | 1 (2) | 1 (1)
Hypotension (Cardiac disorders) | 0 (0) | 1 (1)
Pain in the face (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dry nose (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Headache (General disorders) | 0 (0) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-28): https://cdn.clinicaltrials.gov/large-docs/26/NCT04716426/Prot_SAP_000.pdf